CLINICAL TRIAL: NCT02418559
Title: A Double-Blind, Placebo-Controlled, Randomized, Single Ascending Dose Study to Investigate Safety, Tolerability, and Pharmacokinetics of JNJ-63623872 in Healthy Japanese Adult Subjects
Brief Title: A Study to Investigate Safety, Tolerability, and Pharmacokinetics of JNJ-63623872 in Healthy Japanese Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Infectious Diseases BVBA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR106762; 2015-000247-16 (EudraCT Number); 63623872FLZ1008 (Other: Janssen Infectious Diseases BVBA)
Record Dates: First submitted 2015-04-13; First posted 2015-04-16 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
Keywords: Healthy; JNJ-63623872; Japanese Adult Participants
MeSH Terms: interventions — pimodivir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- JNJ-63623872 (300 mg) or Placebo (Experimental): Participants will receive JNJ-63623872 300 milligram (mg) or placebo tablet orally once on Day 1 under fasted conditions.
  Interventions: Drug: JNJ-63623872 (300 mg); Drug: Placebo
- JNJ-63623872 (600 mg) or Placebo (Experimental): Participants will receive JNJ-63623872 600 mg (2*300 mg) or placebo tablet orally once on Day 1 under fasted conditions.
  Interventions: Drug: JNJ-63623872 (600 mg); Drug: Placebo
- JNJ-63623872 (1200 mg) or Placebo (Experimental): Participants will receive JNJ-63623872 1200 mg (4*300 mg) or placebo tablet orally once on Day 1 under fasted conditions.
  Interventions: Drug: JNJ-63623872 (1200 mg); Drug: Placebo

INTERVENTIONS:
Drug: JNJ-63623872 (300 mg) — Participants will receive JNJ-63623872 300 mg tablet orally once on Day 1 under fasted conditions.
  Arms: JNJ-63623872 (300 mg) or Placebo
Drug: JNJ-63623872 (600 mg) — Participants will receive JNJ-63623872 600 mg (2*300 mg) tablet orally once on Day 1 under fasted conditions.
  Arms: JNJ-63623872 (600 mg) or Placebo
Drug: JNJ-63623872 (1200 mg) — Participants will receive JNJ-63623872 1200 mg (4*300 mg) tablet orally once on Day 1 under fasted conditions.
  Arms: JNJ-63623872 (1200 mg) or Placebo
Drug: Placebo — Participants will receive placebo tablet orally once on Day 1 under fasted conditions.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of JNJ-63623872 following oral administration of single ascending dose of JNJ-63623872 in healthy Japanese adult participants.

DETAILED DESCRIPTION:
This is a double-blind (test or experiment in which neither the person giving the treatment nor the patient knows which treatment the patient is receiving), placebo-controlled, randomized (study medication assigned to participants by chance) and single-center study of JNJ-63623872. The duration of study will be approximately 5.5 weeks for each ISO per participant. The study consists of 3 parts: Screening Phase (28 days before study commences on Day 1); double-blind Treatment Phase (single oral dose of JNJ-63623872 or placebo on Day 1 under fasted condition); and Follow up Phase (up to 7-10 days after study drug administration). All the eligible participants will be randomly assigned to 1 of 3 groups. The planned doses will be escalated in a stepwise fashion if the safety and tolerability in the preceding dose is found acceptable. Participants in Group 1 will receive JNJ-63623872 300 milligram (mg) or placebo, Group 2 will receive JNJ-63623872 600 mg or placebo and Group 3 will receive JNJ-63623872 1200 mg or placebo. Study drug will be administered following a 10-hour overnight fast. Blood samples will be collected for evaluation of pharmacokinetics at pre-dose and post-dose of study treatment. Pharmacokinetics of JNJ-63623872 will be evaluated primarily. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Be a Japanese participant who has resided outside Japan for no more than 5 years and whose parents and grandparents are Japanese as determined by participant's verbal report
* Each participant must sign an Informed Consent Form (ICF) indicating that he or she understands the purpose of and procedures required for the study and are willing to participate in the study
* Participant must be willing and able to adhere to the prohibitions and restrictions specified in this protocol
* A female participant must be either:

  1. Not of childbearing potential: postmenopausal [greater than (>) 45 years of age with amenorrhea for at least 2 years, or any age with amenorrhea for at least 6 months and a serum follicle stimulating hormone (FSH) level >40 International Units (IU)/ liter (L) (to be confirmed at Screening for all postmonopausal women)] OR
  2. Permanently sterilized (eg, bilateral tubal occlusion [which includes tubal ligation procedures as consistent with local regulations], hysterectomy, bilateral salpingectomy, bilateral oophorectomy) or otherwise incapable of becoming pregnant, OR c. If of childbearing potential and heterosexually active, practicing an effective method of birth control before entry and agree to continue to use two effective methods of contraception throughout the study and for at least 30 days after receiving the study drug
* A male participant who is sexually active with a woman of childbearing potential must agree to use two effective methods of birth control for 30 days after receiving the study drug, and a male participant must also not donate sperm during the study and for 3 months after receiving the study drug

Exclusion Criteria:

* Participant has a history of current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the Investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Participant with a past history of heart arrhythmias (extrasystoli, tachycardia at rest), history of risk factors for Torsade de Pointes syndrome (eg, hypokalemia, family history of long QT Syndrome)
* Participants with any history of clinically significant skin disease such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, food allergy, or urticaria
* Participants with a history of clinically significant drug allergy such as, but not limited to, sulfonamides and penicillins, or drug allergy diagnosed in previous studies with experimental drugs
* Participant has taken any disallowed therapies as noted in protocol, Pre-study and Concomitant Therapy before the planned study drug

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of JNJ-63623872 | Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72 and 96 hours post-dose
  The Cmax is the maximum observed plasma concentration of JNJ-63623872.
Time to Reach the Maximum Plasma Concentration (Tmax) of JNJ-63623872 | Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72 and 96 hours post-dose
  The Tmax is the time to reach the maximum observed plasma concentration of JNJ-63623872.
Time of Last Measurable Plasma Concentration (Tlast) of JNJ-63623872 | Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72 and 96 hours post-dose
  Time of last measurable (non-below quantification limit [non-BQL]) plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time 0 to Time of the Last Observed Quantifiable Concentration (AUC [0-last]) of JNJ-63623872 | Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72 and 96 hours post-dose
  The AUC (0-last) is the area under the plasma JNJ-63623872 concentration-time curve from time 0 to time of the last observed (non-BQL) quantifiable concentration, calculated by linear-linear trapezoidal summation.
Area Under the Plasma Concentration-Time Curve From 0 to Infinite Time (AUC[0-infinity]) Post Dose of JNJ-63623872 | Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72 and 96 hours post-dose
  The AUC (0-infinity) is the area under the plasma JNJ-63623872 concentration-time curve from time 0 to infinite time, calculated as the sum of AUC (0-last) and C(last)/lambda(z), in which AUC(0-last) is area under the plasma JNJ-63623872 concentration-time curve from time zero to time of the last quantifiable concentration, C(last) is the last observed (non-BQL) quantifiable concentration and lambda(z) is elimination rate constant. Extrapolations of more than 20.00% of the total AUC are reported as approximations.
Percentage of Area Under the Plasma Concentration-Time Curve Obtained by Extrapolation (%AUC[infinity,ex]) | Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72 and 96 hours post-dose
  The %AUC[infinity,ex] is calculated by dividing the difference of AUC(0-infinity) and AUC(0-last) by AUC(0-infinity) and then multiplying by 100, (AUC[0-infinity] - AUC[0-last])*100/AUC[0-infinity].
Elimination Rate Constant (Lambda [z]) of JNJ-63623872 | Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72 and 96 hours post-dose
  The Lambda (z) determined by linear regression of the terminal points of the ln-linear plasma concentration-time curve.
Apparent Terminal Half-life (t[1/2]) of JNJ-63623872 | Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72 and 96 hours post-dose
  The t(1/2) is defined as 0.693/Lambda (z).
Total Apparent Clearance (CL/F) of JNJ-63623872 | Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72 and 96 hours post-dose
  The CL/F is defined as Dose/AUC (0-infinity).
Apparent Volume of Distribution (Vd/F) of JNJ-63623872 | Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72 and 96 hours post-dose
  The Vd/F is defined as Dose/[Lambda (z)*AUC (0-infinity)].

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious AEs | Screening up to follow-up (7-10 days after dose administration)
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Infectious Diseases BVBA Clinical Trial, Study Director — Janssen Infectious Diseases BVBA
Locations (1):
- Harrow, United Kingdom